CLINICAL TRIAL: NCT03304353
Title: The Efficacy of a Self-managed Resistance Training Protocol Versus a Predetermined Resistance Training Protocol in Reducing Pain in Individuals With Plantar Fasciopathy During a 12-week Intervention: a Randomised Controlled Superiority Trial
Brief Title: Efficacy of a Self-managed Versus a Predetermined Resistance Training Protocol in Reducing Pain in Individuals With Plantar Fasciopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Henrik Riel, PhD Student, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20170051
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Plantar Fasciopathy
Keywords: Plantar heel pain; Resistance training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-managed protocol (Experimental)
  Interventions: Other: Self-managed protocol
- Predetermined protocol (Active Comparator)
  Interventions: Other: Predetermined protocol

INTERVENTIONS:
Other: Self-managed protocol — Participants will be asked to complete a heel raise standing with the forefoot on a step. The toes are maximally dorsi flexed by placing a towel underneath them. The participant is instructed to perform a heel raise to maximal plantar flexion in the ankle joint and afterwards to lower the heel to maximal dorsiflexion. Supporting oneself for balance by placing the hands on a wall or a rail is allowed.
  The participants in the self-managed group are instructed in performing the exercise with a load as heavy as possible but no higher than 8RM and for as many sets as possible every other day.
  Arms: Self-managed protocol
Other: Predetermined protocol — Participants will be asked to complete a heel raise standing with the forefoot on a step. The toes are maximally dorsi flexed by placing a towel underneath them. The participant is instructed to perform a heel raise to maximal plantar flexion in the ankle joint and afterwards to lower the heel to maximal dorsiflexion. Supporting oneself for balance by placing the hands on a wall or a rail is allowed.
  The participants in the predetermined group are instructed in performing the exercise at a 12RM for three sets during week 1 and 2, at a 10RM for four sets during week 3 and 4, and at an 8RM for five sets from week 5 and onwards.
  Arms: Predetermined protocol

SUMMARY:
The purpose of this trial is to investigate whether a self-managed resistance training protocol is more effective than a predetermined resistance training protocol in improving the Foot Health Status Questionnaire pain domain score in individuals with plantar fasciopathy after a 12-week intervention.

DETAILED DESCRIPTION:
This trial will be designed as a randomised, participant-blinded, superiority trial, with a 2-group parallel design to be conducted in Denmark. Reporting of the trial will follow CONSORT guidelines for reporting non-pharmacologic treatments and TIDieR for intervention description. Reporting of the protocol will follow the SPIRIT statement. The planning of the trial was done in accordance with the PREPARE Trial guide (25).

In addition to the exercises, both groups receive patient education on their condition. They will be informed about what is known about the condition in terms of risk factors and aetiology, the pathology, activity modification, and the rationale for why their specific exercise programme (self-managed or predetermined) could lead to recovery. The participants of the predetermined group will be informed that this specific exercise and exercise programme has been found to be superior to stretching but it is important to follow the protocol as closely as possible. The participants of the self-managed group will be informed that this specific exercise has been found to be superior to stretching but based on previous research of other tendinopathies we believe that doing the exercise as heavy as possible but not heavier than 8RM and with as many sets as possible will increase the odds of recovery. Both groups are told that compliance to their protocol is very important and that compliance to the exercises are associated with their recovery. They are also informed about other types of evidence-based treatments however, they are asked to refrain from seeking other treatments during the course of the study. A silicone heel cup will be given to all participants. If the participant already uses an insole or any other type of foot orthosis they will be allowed to continue wearing this if they do not want to use the heel cup.

All statistical analyses will be performed according to a pre-established analysis plan in consultation with a statistician. STATA ver. 14 will be used as statistical software. The primary intention-to-treat analysis will test the between-group difference in the FHSQ pain domain at the 12-week follow-up. In addition to this, between-group comparisons of the other FHSQ domains, PSEQ, IPAQ, and plantar fascia thickness will be performed using a repeated measures ANCOVA with the outcome as the dependent variable, time (baseline, 4 weeks and 12 weeks) as the within-subjects factor, group allocation as the between-subjects factor and the baseline value as the covariate. If any interactions are found, post hoc Bonferroni adjustments for multiple comparisons will be made. The between-group difference in time to PASS among participants who report PASS, and the number of training sessions performed during the trial using independent t-tests. The relative risk (RR) will be calculated for the dichotomized GROC to determine the probability of being improved and for the dichotomized PASS (Yes/No) to determine the probability of achieving a satisfactory result within the 12 weeks of intervention. The difference in mean training sessions performed per week from before to after PASS among participants who report PASS no later than during week 11 of the intervention will be investigated using a paired t-test. The number needed to treat will be calculated as 1/risk difference for the primary outcome. The association between the PSEQ score and compliance will be investigated using Pearson's correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* History of inferior heel pain for at least three months before enrolment
* Pain on palpation of the medial calcaneal tubercle or the proximal plantar fascia
* Thickness of the plantar fascia of 4.0 mm or greater
* Mean heel pain of ≥ 20 mm on a 100 mm VAS [0mm = no pain, 100mm = worst pain imaginable] during the past week

Exclusion Criteria:

* Below 18 years of age
* History of inflammatory systemic diseases
* Pain or stiffness in the 1st metatarsophalangeal joint to an extent where the exercises cannot be performed
* Prior heel surgery
* Pregnancy
* Pain medication
* Corticosteroid injection for plantar fasciopathy within the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Change in Foot Health Status Questionnaire pain domain | At baseline and at the 4- and 12-week follow-ups.
  The Foot Health Status Questionnaire is a self-report questionnaire ranging from 0 (poor foot health) to 100 (optimum foot health) that assesses multiple dimensions of foot health and function. A Danish translation of the original questionnaire will be used. The translation was made using a dual panel approach.

SECONDARY OUTCOMES:
Change in Foot Health Status Questionnaire function domain | At baseline and at the 4- and 12-week follow-ups.
  Ranging from 0 (poor foot health) to 100 (optimum foot health)
Change in Foot Health Status Questionnaire footwear domain | At baseline and at the 4- and 12-week follow-ups.
  Ranging from 0 (poor foot health) to 100 (optimum foot health)
Change in Foot Health Status Questionnaire general foot health domain | At baseline and at the 4- and 12-week follow-ups.
  Ranging from 0 (poor foot health) to 100 (optimum foot health)
Global Rating of Change | At the 12-week follow-up.
  This will be used to measure the participants' self-reported recovery on a 7-point Likert scale ranging from "much improved" to "much worse". Participants are categorised as improved if they rate themselves as "much improved" or "improved" (category 6-7) and categorised as not improved if they rate themselves from "slightly improved" to "much worse" (category 1-5).
Change in plantar fascia thickness | At baseline and at the 4- and 12-week follow-ups.
  Measured in millimeters using ultrasonography
Time to Patient Acceptable Symptom State | From 0 to 12 weeks.
  This will be used as a measure of when the participant achieves a self-reported satisfactory result and is therefore not necessarily a measure of complete recovery. After the participant has reported PASS he or she is still instructed to continue performing the exercise as prescribed.
Change in Pain Self-Efficacy Questionnaire score | At baseline and at the 4- and 12-week follow-ups.
  The Pain Self-Efficacy Questionnaire ranges from 0 (not at all confident) to 60 (completely confident) with lower scores indicating lower self-efficacy. A Danish translation of the original questionnaire, which has been validated in a Danish chronic pain population, will be used.
Change in physical activity level | At baseline and at the 4- and 12-week follow-ups.
  This will be measured using the International Physical Activity Questionnaire short form (IPAQ). A Danish translation of the original questionnaire will be used. The IPAQ is the most commonly used questionnaire for measuring physical activity among adults and consists of 9 items that provide information on the time spent performing vigorous and moderate activities, the time spent walking, and time spent sedentary during the past week. The IPAQ gives an estimate of the total weekly physical activity measured in MET-minutes per week and total minutes spent sitting

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Riel, M.Sc., Principal Investigator — Research Unit for General Practice in Aalborg, Department of Clinical Medicine, Aalborg University
Locations (1):
- Research Unit for General Practice, Aalborg, Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Riel H, Jensen MB, Olesen JL, Vicenzino B, Rathleff MS. Self-dosed and pre-determined progressive heavy-slow resistance training have similar effects in people with plantar fasciopathy: a randomised trial. J Physiother. 2019 Jul;65(3):144-151. doi: 10.1016/j.jphys.2019.05.011. Epub 2019 Jun 13. PMID 31204294

DOCUMENTS (1):
  • Study Protocol (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03304353/Prot_000.pdf